CLINICAL TRIAL: NCT02649088
Title: Sublingual Microcirculation Monitoring in ICU
Acronym: MICRODAIMON
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Associate Professor, Università Politecnica delle Marche
Other Study IDs: 212639
Record Dates: First submitted 2015-12-23; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Critical Illness
Keywords: microcirculation; tissue oxygenation; outcome
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Microscan — It allows to look at sublingual microcirculation
Device: NIRS from Hutchinson — It allows to monitor tissue oxygen saturation

SUMMARY:
Prospective observational study designed to implement a daily monitoring of microcirculation and tissue oxygenation in all critically ill patients admitted to the ICU in the period of nine months, in order to assess the prevalence of microvascular perfusion abnormalities and their relation to: outcomes, underlying disease, hospital stay, clinical-laboratory and hemodynamic parameters commonly measured, indices of clinical severity and predictors of mortality , therapeutic interventions that are part of routine clinical practice (fluids, sedation, vasopressors, inotropes, anticoagulants, renal replacement therapy, blood transfusion). The study also includes the evaluation of sublingual microcirculation and tissue oxygenation in 30 healthy volunteers to compare normal and pathological conditions. Within the first 12 hours after admission to ICU and every 24 hours for the duration of hospitalization, the following evaluations will be made: -study of sublingual microcirculation using sidestream dark field (SDF) imaging, muscle tissue oxygenation using near infrared spectroscopy (NIRS). The data will be analyzed to test correlation between the outcome of patients admitted in ICU and microcirculatory parameters.

DETAILED DESCRIPTION:
The aim of this study is to daily assess microcirculation and tissue oxygenation in all critically ill patients admitted to the ICU during a period of nine months, in order to assess the prevalence of microvascular perfusion abnormalities and their relation to: outcomes, underlying disease, duration of hospitalization, clinical-laboratory and hemodynamic parameters commonly measured, indices of clinical severity and predictors of mortality (SAPS II , APACHE II , SOFA score , PIRO score ), therapeutic interventions are part of common clinical practice (fluids, sedation, vasopressors, inotropes, anticoagulants, renal replacement therapy, blood transfusion). In order to implement a comparison between normal and pathological conditions, sublingual microcirculation and tissue oxygenation will be assessed "una tantum" in 35 healthy volunteers.

STATISTICAL ANALYSIS: Descriptive statistics will be used to describe the population of patients recruited. The prevalence of Microcirculatory abnormalities will be assessed in the general population and in distinct patient subgroups based on the underlying disease. Receiver operator curve (ROC) Curves will be used to determine cut-off values for Microcirculatory variabile s related to morbidity and mortality. It will be assessed the correlation between variables and Microcirculatory: hemodynamic parameters and laboratory, length of stay in ICU/hospital, APACHE II, SAPS II, mortality, SOFA, PIRO score (the latter for septic patients). Multivariate analysis will be used to assess the association between Microcirculatory alterations and other variables. Microcirculatory differences among various subgroups (differentiated by outcome, underlying disease, severity indices, therapies; if sepsis: site of infection) will be assessed using t-test (for normally distributed variables) or with non-parametric tests for not normally distributed variables.

MATERIAL AND METHODS: ICU is divided into three subunits: Respiratory ICU, Medical ICU and Trauma ICU with 4 beds each. All patients admitted in each subunit have been daily monitored from the admission until the discharge for a period of 3 months. The subunits will be included in the study not at the same time but sequentially so that the total period for monitoring will be of 9 months. In order to implement a comparison between normal and pathological conditions, sublingual microcirculation and tissue oxygenation are evaluated in 35 healthy volunteers, which will be adequately informed of the aims and methods of the study and will give their written consent. The comparison between healthy volunteers and patients is necessary because the normal values for Microcirculatory parameters have not yet been established. It should be noted that all healthy volunteers will be recruited within the current staff of ICU and measurements will be performed only once. Within the first 12 hours after admission and every 24 hours for the duration of hospitalization, sublingual microcirculation is evaluated by using the technique of sidestream dark field (SDF) imaging currently used in our Department (Microscan, Microvision Medical, Amsterdam, The Netherlands). Contextually sublingual microcirculation study, tissue oxygenation will be evaluated using near infrared spectroscopy (NIRS), already in widespread use in our clinical practice (InSpectra ™ Model 650; Hutchinson Technology Inc., Hutchinson, MN, USA, nr. inventory status: 15852). For each patient the following data will be collected: age, sex, diagnosis, APACHE II, SAPS II, past medical history (arterial hypertension, diabetes mellitus, chronic renal failure, cardiovascular, cerebrovascular, liver cirrhosis, immune deficiencies, therapy with beta-blockers, Nitro), results of microbiological tests, SOFA score, PIRO score (septic patients), length of stay in hospital and in intensive care, outcome. Every day, parameters routinely assessed in clinical practice will be collected: body temperature, heart rate, mean arterial pressure, hemodynamic parameters (where femoral catheter already exists Cardiac index (CI), Intrathoracic blood volume ( ITBVI), EVLWI), blood gas analysis parameters (pH, PaO2, PaCO2, BE, PaO2/FiO2, lactates); fluid balance, diuresis; complete blood count (hemoglobin, hematocrit, WBC, RBC, PLT), creatinine, glucose (from arterial blood drawn for abgs-analysis), total bilirubin, PCR, Procalcitonin (if any), INR, PT, PTT, Fibrinogen; therapies: analgo-sedation, inotropes, vasopressors, blood transfusion, fluids. EVALUATION OF MICROCIRCULATION After removing any secretions with gauze, the probe will be gently applied to the sublingual mucosa without exerting excessive pressure. At each timepoint, videos from 3-5 different sites of a minimum duration of 10 seconds each will record. After assigning a random number, the images will be analyzed with a dedicated software and, in accordance with the criteria established in a roundtable of experts in 2007 [17], laid down the following variables: De Backer score, Total Vessel Density (TVD) and hearts Perfused Vessel Density (PVD), which indexes the density of perfused vessels; Microvascular Flow Index (MFI) and Proportion of Perfused Vessels (PPV), perfusion quality indices; Flow Heterogeneity Index (HI), index of homogeneity of flow distribution. The images will also be analyzed using the ICU GlycoCheck (Maastricht University Medical Center, Maastricht, The Netherlands, www.glycocheck.com) to get the value of the Perfused Boundary Region (PBR, micron), which represents the thickness of the permeable of glycocalyx that allows the penetration of erythrocytes, damage index of glycocalyx. TISSUE OXYGENATION ASSESSMENT Tissue oxygenation is assessed at rest and during a test of forearm vascular occlusion. NIRS probe will be placed at the level of the thenar eminence and the cuff of a sphygmomanometer around the forearm; After 3 minutes the signal stabilisation, the cuff is inflated to a pressure 40 mmHg higher than the patient's systolic to block the flow of blood. You will wait so that the descent of StO2 until 40% prior to deflate the cuff. The rate of descent of StO2 ischemic phase (StO2 downslope) is an indication of extraction and consumption of O2; the ascent rate during reperfusion (StO2 upslope), along with the area under the curve during the next stage of reactive hyperemia (AUC StO2), is an indication of the reactivity of the micro-circulation. It should be noted that vascular occlusion testing is absolutely harmless, because the phase of ischemia is too short (usually 2-3 minutes at most) in order to cause any ischemic damage to the tissues of the limb. The Tissue Hemoglobin Index (THI), reflecting the contents of Hb in volume of muscle tissues assessed by the probe, depends not only by blood levels of Hb, but also the density of capillaries perfused.

Finally glycocalyx assessment will be done and it will compared among volunteers, septic critically ill patients and non-septic critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted in ICU

Exclusion Criteria:

* age <18
* expected ICU length of stay <24 hrs
* any conditions that preclude sublingual microcirculatory evaluation (e.g. facial trauma)
* readmitted patients previously enrolled in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in perfused vessel density and 90 days mortality from ICU admission | 90 days
  The perfused vessel density (PVD) is defined as the quantity (mm/mmq) of microcirculatory vessels which have a good flow and it is calculated using a dedicated software described elsewhere.
Correlation between changes in StO2 upload and 90 days mortality from ICU admission | 90 days
  During vascular occlusion test, the changes of StO2 and StO2 values can divided into 3 epoch; Desaturation (StO2 download), Reoxygenation (StO2 upload), and Reactive hyperemia. After data collection, the rate of desaturation and reoxygenation are calculated.

SECONDARY OUTCOMES:
Correlation between Perfused vessel density and central venous saturation | Study frame: nine months
  The perfused vessel density (PVD) is defined as the quantity (mm/mmq) of microcirculatory vessels which have a good flow and it is calculated using a dedicated software described elsewhere. Central Venous Saturation is measured from a blood sample from a central venous catheter.
Correlation between Perfused vessel density and blood lactate | Study frame: nine months
Correlation between Perfused vessel density and ICU length of stay | Study frame: nine months
Correlation between Perfused vessel density and hospital length of stay | Study frame: nine months
Correlation between Perfused vessel density and SOFA score | Study frame: nine months
Glycocalyx assessment among volunteers, septic and non septic critically ill patients | Study frame: nine months
  Glycocalyx is indirectly measured using a dedicated software as described in a previous paper

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- University ICU, AOU Ospedali Riuniti Ancona, Torrette Di Ancona, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scorcella C, Damiani E, Domizi R, Pierantozzi S, Tondi S, Carsetti A, Ciucani S, Monaldi V, Rogani M, Marini B, Adrario E, Romano R, Ince C, Boerma EC, Donati A. MicroDAIMON study: Microcirculatory DAIly MONitoring in critically ill patients: a prospective observational study. Ann Intensive Care. 2018 May 15;8(1):64. doi: 10.1186/s13613-018-0411-9. PMID 29766322
- [Derived] Donati A, Damiani E, Domizi R, Scorcella C, Carsetti A, Tondi S, Monaldi V, Adrario E, Romano R, Pelaia P, Singer M. Near-infrared spectroscopy for assessing tissue oxygenation and microvascular reactivity in critically ill patients: a prospective observational study. Crit Care. 2016 Oct 1;20(1):311. doi: 10.1186/s13054-016-1500-5. PMID 27716370